CLINICAL TRIAL: NCT03364530
Title: Hepatic Arterial Infusion of Gemcitabine-oxaliplatin for Second-line Therapy in Non-metastatic Unresectable Intra-hepatic Cholangiocarcinoma: a Multicentric Single-arm Phase II Study
Brief Title: Hepatic Arterial Infusion of Gemcitabine-oxaliplatin for Second-line Therapy in Non-metastatic Unresectable Intra-hepatic Cholangiocarcinoma
Acronym: GEMOXIA-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL17_0025; UF 9794 (Other: Montpellier University Hospital)
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cholangiocarcinoma Non-resectable; Non-metastatic
MeSH Terms: interventions — gemcitabine-oxaliplatin regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine-Oxaliplatin Regimen (Other)
  Interventions: Drug: Gemcitabine-Oxaliplatin Regimen; Procedure: Hepatic intra arterial chemotherapy

INTERVENTIONS:
Drug: Gemcitabine-Oxaliplatin Regimen — Vascularisation of hepatic tumors is almost exclusively provided by the hepatic artery.
  Gemcitabine and oxaliplatin have a high rate of hepatic extraction during the first passage, thus allowing the drugs to reach high intra-tumoral concentrations with low systemic toxicity.
Procedure: Hepatic intra arterial chemotherapy — The implantation of a hepatic arterial catheter has now been mastered by interventional radiologists and makes it possible to increase the intra-tumoral concentration of the drugs and probably to limit their systemic toxicity.
  Very recently, we have reported that this combination in progressive IHC following systemic gemcitabine/oxaliplatin has led to partial responses and allowed certain patients to benefit from curative treatment.
  This suggests that the intra-arterial approach increases the efficacy of these 2 drugs. For locally-advanced IHC, such a loco-regional approach is worth exploring in this poor-prognosis tumor.

SUMMARY:
We hypothesized that intra-arterial gemcitabine/oxaliplatin administered as second-line treatment could strongly improve objective response rate at 4 months after inclusion in patient with non-metastatic unresectable intra-hepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Cholangiocarcinomas are rare tumors with an extremely poor prognosis. The best therapeutic option (i.e. resection) can only be done in 20% of cases. Combinations of gemcitabine/platinum compounds were identified as the new standard first-line therapy

For patients with hepatic-only disease, therapy intensification using Intra-Arterial (IA) chemotherapy could be an attractive option since:

* Vascularisation of hepatic tumors is almost exclusively provided by the hepatic artery.
* Gemcitabine and oxaliplatin have a high rate of hepatic extraction during the first passage, thus allowing the drugs to reach high intra-tumoral concentrations with low systemic toxicity.
* The plasma concentration of gemcitabine after IA injection is 1/7th of that observed following Intra-Venous (IV) injection. No grade 3-4 toxicity has been observed in doses <1400mg/m².
* Phase I and I/II studies have shown dose-limiting toxicity between 150-175mg/m² for IA oxaliplatin every 3 weeks.
* We reported (Ghiringhelli, Chemotherapy 2013) in 12 patients with progressive intra-hepatic cholangiocarcinoma after IV gemcitabine/oxaliplatin, a partial response in 8 cases (stability in 3 cases) after IA gemcitabine/oxaliplatin. Among them, two were resected (R0) and three were treated by stereotactic radiation therapy).

Hepatic IA chemotherapy has rarely been used for the treatment of intra-hepatic cholangiocarcinoma (IHC), essentially in case-reports from Asia and in a few case-series that have mainly used IA monotherapy. The implantation of a hepatic arterial catheter has now been mastered by interventional radiologists and makes it possible to increase the intra-tumoral concentration of the drugs and probably to limit their systemic toxicity.

Very recently, we have reported that this combination in progressive IHC following systemic gemcitabine/oxaliplatin has led to partial responses and allowed certain patients to benefit from curative treatment.

This suggests that the intra-arterial approach increases the efficacy of these 2 drugs. For locally-advanced IHC, such a loco-regional approach is worth exploring in this poor-prognosis tumor, especially since so far 1) there is insufficient evidence to recommend a second-line chemotherapy schedule in this tumor and 2) targeted therapies have demonstrated no survival benefit over systemic chemotherapy alone.

It is a multicenter single-arm phase II trial aiming to determine the objective response rate 4 months after inclusion following IA gemcitabine / oxaliplatin administered as second-line treatment in patients with non-metastatic unresectable intra-hepatic cholangiocarcinoma.

It will be the first French phase II trial for 2nd line treatment in intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven intrahepatic cholangiocarcinoma previously treated by first-line systemic therapy
* Absence of extra-hepatic metastasis or peritoneal carcinomatosis (as demonstrated by CT-scan)
* General health status : World Health Organization Performance Status = 0, 1
* Estimated life expectancy > 3 months
* Disease that is not suitable for resection with a curative intent, as validated by a multidisciplinary committee with at least one senior hepatic surgeon
* At least one measurable lesion according to RECIST 1.1 criteria
* Platelets ≥100,000/mm3, polynuclear neutrophils ≥ 2000/mm3 , hemoglobin 9g/dL (even transfused patients can be included)
* Creatininemia < 1.5 mol/L
* Creatinine clearance > 30 mL/min
* Bilirubinemia ≤2 N (after biliary drainage if necessary)
* Aspartate and Alanine Transaminase ≤ 5 mol/L
* Reference hepatic MRI (according to the foreseen protocol) done during the 30 days preceding the 1st cycle of treatment
* Written informed consent
* National health insurance cover

Exclusion Criteria:

* Patients with cholangiocarcinoma of the gallbladder or common bile duct or those with hepatocholangiocarcinoma or a Klatskin tumor
* Patients who are eligible for surgical resection or liver transplantation
* Extra-hepatic metastases (Pulmonary micronodules <7mm without uptake on positron emission tomography are not a contra-indication)
* Presence of clinical ascites
* History of intra-arterial therapy or more than one line of systemic treatment
* Contra-indication or grade 3-4 allergy to any of the treatment drugs Gemcitabine, Oxaliplatin (notably myelosuppression developped before the beginning of the first cycle of therapy, peripheral sensory neuropathy before the first cycle of therapy, severe renal failure)
* Grade 2 peripheral neuropathy
* Ongoing participation or participation within the 21 days prior to inclusion in the study in another therapeutic trial with an experimental drug
* Concomitant systemic treatment with immunotherapy, chemotherapy or hormone therapy
* Serious non-stabilized disease, active uncontrolled infection or other serious underlying disorder likely to prevent the patient from receiving the treatment
* Pregnancy (beta-human chorionic gonadotropin positive), breast-feeding or the absence of effective contraception for women of child-bearing age
* Another cancer in the 5 years preceding or at the time of inclusion in the trial (except for in situ cervical cancer or basal cell carcinoma of the skin)
* Allergy or contra-indication to iodine contrast agents (thyrotoxicosis, allergy to the active substance or excipients)
* Treatment with anticoagulants (heparin or AVK) that cannot be interrupted for 12 hours
* Treatment with anti-platelets that cannot be interrupted for 5 days for aspirin or Plavix.
* Contra-indication for use of an intra-arterial approach (severe arteriopathy)
* Legal incapacity (persons in custody or under guardianship)
* Deprived of liberty Subject (by judicial or administrative decision)
* Impossibility to sign the informed consent document or to adhere to the medical follow-up of the trial for geographical, social or psychological reasons
* Contraindication for the MRI : Pacemaker or neurosensorial stimulator or implantable defibrillator, cochlear implant, ferromagnetic foreign body similar to the nervous structure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 4 months after inclusion
  The primary outcome is to evaluate the objective response rate (complete or partial response) 4 months after inclusion using RECIST 1.1 evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Boris GUIU, Principal Investigator — Montpellier University Hospital
Locations (7):
- France (7):
  - Amiens University Hospital, Amiens
  - Angers University Hospital, Angers
  - Bordeaux University Hospital, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Uhmontpellier, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No